CLINICAL TRIAL: NCT02963207
Title: Prospective Randomised Study Comparing Modified Sano's (MS) Classification and NBI International Colorectal Endoscopic (NICE) for Differentiating Colorectal Lesions
Brief Title: MS Versus NICE for Colorectal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lyell McEwin Hospital (Other Government)
Collaborators: University of Adelaide (Other)
Responsible Party: Principal Investigator, Leonardo Zorron Cheng Tao Pu, Research Fellow, Lyell McEwin Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2008128
Record Dates: First submitted 2016-11-06; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Neoplasms; Colorectal Polyp
Keywords: colorectal polyp; colorectal lesion; Modified Sano's Classification; NICE classification; NBI; PIVI guidelines; SSA/P; sessile serrated adenoma; sessile serrated polyp
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified Sano's Classification (Experimental): Modified Sano's Classification as described by Singh et al. 2013
  Interventions: Other: Modified Sano's classification
- NICE classification (Active Comparator): NBI International Colorectal Endoscopic Classification as described by Hewett et al. 2012
  Interventions: Other: NICE classification

INTERVENTIONS:
Other: Modified Sano's classification — Set of characteristics described by Singh et al. 2013 to evaluate colorectal lesions.
  Other Names: MS classification
  Arms: Modified Sano's Classification
Other: NICE classification — Set of characteristics described by Hewett et al. 2012 to evaluate colorectal lesions.
  Other Names: NBI International Colorectal Endoscopic Classification
  Arms: NICE classification

SUMMARY:
OBJECTIVE: Our study aimed to compare a recently-developed endoscopic classification with an established one for colorectal lesions in a randomised trial between 2013 and 2015.

DETAILED DESCRIPTION:
OBJECTIVE: Current practice requires histopathological assessment to confirm diagnosis for colorectal lesions detected at colonoscopy. Advances in endoscopic imaging contribute for real-time diagnosis which, apart from being cost and time-saving, also guides decision-making and reduces risks. Our study aimed to compare a recently-developed endoscopic classification with an established one.

DESIGN: The modified Sano's classification (MS) was compared to the Narrow Band Imaging (NBI) International Colorectal Endoscopic classification (NICE) in a randomised trial between 2013 and 2015. An experimented endoscopist classified each polyp, what was compared to histopathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the Endoscopy Unit for a colonoscopy
* Patients over 18 years-old
* Patients or their caregivers that have understanding of the procedure and that have signed the consent form for the study

Exclusion Criteria:

* Patients without colorectal polyps
* Patients with poor bowel preparation
* Patients that do not agree with or withdraw the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Accuracy measures in comparison to the final histopathology in regards to polyps' subtype (neoplastic versus non-neoplastic) | After two weeks of the colonoscopy
  Comparison of NICE or MS with the final histopathology in regards to polyps' subtype (i.e. non-neoplastic = Hyperplastic Polyp (HP) and neoplastic = Sessile Serrated Adenoma/Polyp (SSA/P), Adenomatous Polyp (AP), Traditional Serrated Adenoma (TSA), superficial cancer and invasive cancer)
Accuracy measures in comparison to the final histopathology in regards to polyps' invasiveness | After two weeks of the colonoscopy
  Comparison of NICE or MS with the final histopathology in regards to invasiveness (SSA/P, AP, TSA or superficial cancer versus invasive cancer)
Accuracy measures in comparison to the final histopathology in regards to polyps' subtype (SSA/P versus non-SSA/P) | After two weeks of the colonoscopy
  Comparison of MS with the final histopathology in regards to SSA/P (SSA/P versus non-SSA/P)

SECONDARY OUTCOMES:
Accuracy in regards to negative predictive value of diminutive distal colorectal polyps | After two weeks of the colonoscopy
  Comparison of NICE or MS with the final histopathology in regards to <5 mm distal to the sigmoid polyps (NPV for HPs - according to the PIVI guidelines)
Agreement in predicting post-colonoscopy surveillance interval with final histopathology | Immediately after the colonoscopy (endoscopic) and 2 weeks after (histopathology)
  Comparison of NICE or MS with the final histopathology in regards to prediction of surveillance interval (according to the PIVI guidelines)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo ZC Pu, MD, MSc, Principal Investigator — The Lyell McEwin and The University of Adelaide

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh R, Jayanna M, Navadgi S, Ruszkiewicz A, Saito Y, Uedo N. Narrow-band imaging with dual focus magnification in differentiating colorectal neoplasia. Dig Endosc. 2013 May;25 Suppl 2:16-20. doi: 10.1111/den.12075. PMID 23617643
- [Background] Hewett DG, Kaltenbach T, Sano Y, Tanaka S, Saunders BP, Ponchon T, Soetikno R, Rex DK. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology. 2012 Sep;143(3):599-607.e1. doi: 10.1053/j.gastro.2012.05.006. Epub 2012 May 15. PMID 22609383